CLINICAL TRIAL: NCT05187195
Title: The Effects of Two Different Tele-rehabilitation Interventions on Physical Parameters and Activities of Daily Living in People With Parkinson's Disease
Brief Title: The Effects of Tele-rehabilitation Interventions in Parkinson's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Elif Yılmaz, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUC-2021/48
Record Dates: First submitted 2021-12-24; First posted 2022-01-11 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Parkinson Disease
Keywords: Telerehabilitation; Physical Therapy Modalities; Nervous System Diseases; Home-based; Physiotherapy
MeSH Terms: conditions — Parkinson Disease; Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation-video group (Experimental): This group will perform their exercises with prepared personalized exercise videos through the telerehabilitation system 3 days a week for 8 weeks.
  Interventions: Other: Home-based telerehabilitation with exercise videos
- Telerehabilitation-brochure group (Experimental): This group will perform exercises with personalized exercise brochures defined through the telerehabilitation system 3 days a week for 8 weeks.
  Interventions: Other: Exercise brochure

INTERVENTIONS:
Other: Home-based telerehabilitation with exercise videos — Balance, walking, strengthening, posture videos etc. taken in different positions will be uploaded to the telerehabilitation system. A personalized exercise program will be created from these exercises. This program will be defined to the account of the patient and the follow-up of the person will be carried out through the system.
  Arms: Telerehabilitation-video group
Other: Exercise brochure — Photos and explanations of exercises taken in different positions such as balance, walking, strengthening, posture etc. will be uploaded to the telerehabilitation system. A personalized exercise brochure will be created from these exercises. This program will be defined for the patient's account and the patient will be asked to follow the exercises with this brochure.
  Arms: Telerehabilitation-brochure group

SUMMARY:
Parkinson's Disease (PD) is the most common neurodegenerative movement disorder. The main motor symptoms of PD are tremor, rigidity, bradykinesia, and postural instability. Current treatments of the disease provide control of motor symptoms but do not change its development. Parkinson's patients should receive regular rehabilitation as part of their treatment. Telerehabilitation (TR) practices and studies examining the effectiveness of these practices are needed in order to reduce the impact of the current pandemic period and environmental and personal causes in accessing rehabilitation services.

In this thesis, in order to examine the effects of two different TR methods on physical parameters and activities of daily living in Parkinson's patients, Parkinson's patients who are eligible the inclusion criteria will be randomized according to the row of application and divided into 2 groups. Evaluations to determine the functionality, activities of daily living, falling activity, quality of life and fatigue level will be applied both groups. One group will be applied video exercise program prepared individually via TR system, and the other group will receive an exercise brochure via the TR system and patients will be asked to do the exercises 3 days a week for 8 weeks. Then the initial evaluations will be repeated. It is aimed to increase functional capacity, independence in daily living activities and quality of life, and reduce the number of falls and fatigue levels with exercise training to be applied to people with Parkinson's.

Investigators think that present study not only will contribute to the field of TR applications in PD, but also will provide access to rehabilitation services and help control symptoms of Parkinson's patients who cannot go to hospital, rehabilitation centers and cannot access rehabilitation services at home.

Hypotheses:

H0-TR applications have no effect on the level of independence in physical parameters and activities of daily living in individuals with PD.

H1-TR applications have positive effects on physical parameters and independence in activities of daily living in individuals with PD.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Parkinson's disease at least 1 year ago by a neurologist
* Hoehn and Yahr score ≤3
* Have an internet infrastructure where the system can be accessed at home
* Not participating in a standardized physiotherapy program in the last 3 months

Exclusion Criteria:

* Presence of blurred or low vision problems
* Hearing and speech impairment affecting participation in the system
* Epilepsy
* Presence of pregnancy
* Having any cognitive problems that prevent using the system

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-11-14 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Single Leg Stance Test - SLS (The change between the initial value and value after 2 months will be evaluated) | Baseline and end of weeks 8
  It is a functional assessment test that measures the patient's standing balance on one leg. It is applied for both legs of the patient with eyes open and closed. In Parkinson's disease, standing for less than 10 seconds is associated with balance problems and the risk of falling. Standing for a long time indicates better function. The test maintains for a maximum of 1 minute.
Five Times Sit to Stance Test - 5XSST (The change between the initial value and value after 2 months will be evaluated) | Baseline and end of weeks 8
  This test assesses functional lower extremity strength, transfer, balance, and fall risk. The time the patient sits and stands up from the chair 5 time is recorded. Lasting longer than 16 seconds is associated with the risk of falling in Parkinson's patients. Completing the movement in less time indicates better function.
Romberg Test - RT (The change between the initial value and value after 2 months will be evaluated) | Baseline and end of weeks 8
  The patient's standing time is recorded in an upright position with her feet open at shoulder level and arms free at the side of the body, with her eyes open and then closed, without losing her balance. If the patient cannot stand with his eyes closed, the test is considered positive, and if the patient can stand with his eyes closed, the test is considered negative. The test is continued for a maximum of 60 seconds. Being able to stand longer indicates better function.
Independent Standing Test (The change between the initial value and value after 2 months will be evaluated) | Baseline and end of weeks 8
  It tests the patient's ability to stand in an upright position without any support or assistance, with her feet shoulder width apart and arms free at the side of the body. The patient is expected to be able to stand for 20 seconds. Being able to stand longer indicates better function.
Katz Index of Independence in Activities on Daily Living (The change between the initial value and value after 2 months will be evaluated) | Baseline and end of weeks 8
  It is a scale that measures the patient's ability to perform activities of daily living independently and evaluates the functional status. The patient can get a minimum of 0 points and a maximum of 7 points. Higher score indicates better status.

SECONDARY OUTCOMES:
Modified Falls Efficacy Scale (The change between the initial value and value after 2 months will be evaluated) | Baseline and end of weeks 8
  It is a 14-item scale that measures the patient's confidence in falling. The patient can get a minimum of 0 points and a maximum of 140 points. Higher score indicates better status.
The World Health Organization Quality of Life Instrument, Short Form, Turkish Version (WHOQOL-BREF-TR) (The change between the initial value and value after 2 months will be evaluated) | Baseline and end of weeks 8
  It is a health-related quality of life scale developed by the World Health Organization. A national question was added to Turkish version of the scale in addition to the original version. Each item on the 26-item scale should be evaluated on its own. Scoring is made from 1 to 5. In some questions, 1 indicates a positive situation, while in some questions 5 indicates positive thoughts.
Fatigue Severity Scale (The change between the initial value and value after 2 months will be evaluated) | Baseline and end of weeks 8
  It is a scale that evaluates the severity of fatigue with 9-items that patients can answer on their own. The patient can get a minimum of 9 points and a maximum of 63 points. A lower score indicates better status.
Global Rating of Change Scales | End of weeks 8
  It is a scale that evaluates how much the patient's current condition has changed compared to previous condition. The patient can get a minimum of -5 and a maximum of 5 points. Higher score indicates better status.
System Usability Scale | End of weeks 8
  It is a scale consisting of 10 questions widely used in the literature to evaluate the perceptibility and usability of interactive systems. Each item on the 10-item scale should be evaluated on its own. Scoring is made from 1 to 5. In some questions, 1 indicates a positive situation, while in some questions 5 indicates positive thoughts.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yılmaz, M.Sc, Principal Investigator — Istanbul University- Cerrahpasa Institute of Postgraduate Education; Yonca Zenginler Yazgan, PhD, Study Chair — Istanbul University- Cerrahpasa Faculty of Health Science
Locations (1):
- İstanbul University-Cerrahpasa, Istanbul, Buyukcekmece, Turkey (Türkiye)